CLINICAL TRIAL: NCT02318446
Title: Efficacy Study of Folic Acid Supplementation on Homocysteine Levels in Adolescent Epileptics Taking Antiepileptic Drugs: A Single Blind Randomized Controlled Clinical Trial
Brief Title: Efficacy Study of Folic Acid Supplementation in Adolescent Epileptics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Uma Bhosale, Professor in Department of Pharmacology, SKNMC & GH, Pune-41, Maharashtra University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTRG/E-1/03/ 1210
Record Dates: First submitted 2014-12-10; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
Keywords: Anti-epileptic drugs; Folic acid; Homocysteine
MeSH Terms: conditions — Epilepsy | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Will receive Oral saccharine tablet daily for 1month along with their existing antiepileptic therapy
  Interventions: Drug: Saccharine
- Test group (Experimental): Will receive Oral Folic acid 1mg tablet daily for 1month along with their existing antiepileptic therapy
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Folic Acid — Test group(n= 24) Existing Anti-epileptic Drugs + Oral Folic acid 1mg tablet daily for 1month
  Other Names: Folvite
  Arms: Test group
Drug: Saccharine — Placebo group(n=12) Existing Anti-epileptic Drugs + Oral saccharine 10 mg tablet daily for 1month
  Other Names: Sugar free
  Arms: Control group

SUMMARY:
The present study is planned to study effect of folic acid supplementation on homocysteine levels and CV risk factors such as BP and lipids in adolescent epileptics taking anti-epileptic drugs (AEDs).

DETAILED DESCRIPTION:
Scientific background, significance and impact value of the project:

Homocysteine is a thiol-containing amino acid formed as an intermediate product during the methionine metabolism. Re-methylation pathway recycles Homocysteine back to methionine and requires vitamin B12 and folic acid as cofactors. [1] The concentration of circulating total homocysteine is a sensitive marker of inadequate folate and vitamin B12 status. Elevated homocysteine concentrations are associated with an increased risk for cardiovascular (CV) disease. [2] The total homocysteine level is the lowest in children and an increase with age is higher in male sex. [2] The cutoffs for homocysteine level in adolescent range from 4.3 to 9.9 µmol/l, and hyperhomocysteinemia is defined as homocysteine >10.9 µmol/l. [3] Lower folate and higher homocysteine concentrations may put adolescent on AEDs at special risk for atherosclerosis in their adulthood. [4] This demands early intervention as Asian Indian adolescents are genetically more exposed to cadiovascular disease(CVD) risks, AED therapy is an additional risk for developing future CVDs. Adolescent epileptics on AED have to take it for long time, and homocysteine elevation itself has got epileptogenic potential and can cause the risk developing refractory epilepsy. [5] Literature search reveals several studies depicting role of vitamin B12 in regulation of blood homocysteine levels. [6, 7] However, the studies confirming role of folic acid supplementation in hyperhomocysteinemia and related CV diseases are fewer and scarce in AEDs induced hyperhomocysteinemia. Few studies have reported negative correlation between hyperhomocysteinemia and low folic acid levels in patients on AEDs. [8] At the same time few studies have reported effectiveness of folic acid supplementation to normalize the homocysteine levels. [9] Considering the results of various studies many doctors are now prescribing folic acid along with AEDs, although there is a scarcity of data from India. In this context, the present study is planned to study effect of folic acid supplementation on homocysteine levels and CV risk factors such as BP and lipids in adolescent epileptics taking AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed epileptic patients of either sex with age between 10-19 yrs (<19yrs), coming to the medicine Out Patient /In Patient Departments and undergoing AED therapy for more than 6 months.
* Epileptics with high homocysteine levels i.e. > 10.9 µmol/L (Normal homocysteine levels are 4.3-9.9 µmol/L for male and 3.3-7.2 µmol/L for female adolescent and a high homocysteine concentration is deaned as at least 11.4 µmol/L for male and at least 10.4 µmol/L for female. Gender mean of high homocysteine concentration is 10.9 µmol/L) [5]

Exclusion Criteria:

* Pregnancy and lactation
* Patients with diabetes, Ischemic heart disease (IHD), stroke, malignancy and psychiatric diseases are excluded from study.
* The patients receiving vitamin supplements or who had clinical evidence for an acute illness, renal dysfunction, thyroid dysfunction, chronic inflammatory diseases, inborn errors of homocysteine, cobalamin or folate metabolism, or any other condition known to interfere with homocysteine metabolism will be excluded
* Patients who are already involved in any other trial.
* Patients not willing to fill consent/ assent form are also excluded from study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Decrease in serum homocysteine levels by 2 µmol/l | 1 month

SECONDARY OUTCOMES:
Change in baseline serum lipids | 1 month
  Change in baseline serum lipids following Anti-epileptic therapy will be compared between placebo and test group.
Change in baseline systolic blood pressure | 1 month
  Change in baseline systolic blood pressure will be compared between placebo and test group.

CONTACTS AND LOCATIONS:
Overall Officials: UMA A. BHOSALE, MD, Principal Investigator — Smt. Kashibai Navale Medical College and General Hospital
Locations (1):
- Smt. Kashibai Navale Medical College and General Hospital, Pune, Maharashtra, India

REFERENCES:
- [Background] Hoffer LJ. Homocysteine remethylation and trans-sulfuration. Metabolism. 2004 Nov;53(11):1480-3. doi: 10.1016/j.metabol.2004.06.003. PMID 15536605
- [Background] Selhub J, Miller JW. The pathogenesis of homocysteinemia: interruption of the coordinate regulation by S-adenosylmethionine of the remethylation and transsulfuration of homocysteine. Am J Clin Nutr. 1992 Jan;55(1):131-8. doi: 10.1093/ajcn/55.1.131. PMID 1728812
- [Background] Selhub J, Jacques PF, Rosenberg IH, Rogers G, Bowman BA, Gunter EW, Wright JD, Johnson CL. Serum total homocysteine concentrations in the third National Health and Nutrition Examination Survey (1991-1994): population reference ranges and contribution of vitamin status to high serum concentrations. Ann Intern Med. 1999 Sep 7;131(5):331-9. doi: 10.7326/0003-4819-131-5-199909070-00003. PMID 10475885
- [Background] Osganian SK, Stampfer MJ, Spiegelman D, Rimm E, Cutler JA, Feldman HA, Montgomery DH, Webber LS, Lytle LA, Bausserman L, Nader PR. Distribution of and factors associated with serum homocysteine levels in children: Child and Adolescent Trial for Cardiovascular Health. JAMA. 1999 Apr 7;281(13):1189-96. doi: 10.1001/jama.281.13.1189. PMID 10199428
- [Background] Cheng LS, Prasad AN, Rieder MJ. Relationship between antiepileptic drugs and biological markers affecting long-term cardiovascular function in children and adolescents. Can J Clin Pharmacol. 2010 Winter;17(1):e5-46. Epub 2010 Jan 4. PMID 20051609
- [Background] Sato Y, Ouchi K, Funase Y, Yamauchi K, Aizawa T. Relationship between metformin use, vitamin B12 deficiency, hyperhomocysteinemia and vascular complications in patients with type 2 diabetes. Endocr J. 2013;60(12):1275-80. doi: 10.1507/endocrj.ej13-0332. Epub 2013 Sep 8. PMID 24018893
- [Background] Satyanarayana A, Balakrishna N, Pitla S, Reddy PY, Mudili S, Lopamudra P, Suryanarayana P, Viswanath K, Ayyagari R, Reddy GB. Status of B-vitamins and homocysteine in diabetic retinopathy: association with vitamin-B12 deficiency and hyperhomocysteinemia. PLoS One. 2011;6(11):e26747. doi: 10.1371/journal.pone.0026747. Epub 2011 Nov 1. PMID 22069468
- [Background] Coppola G, Ingrosso D, Operto FF, Signoriello G, Lattanzio F, Barone E, Matera S, Verrotti A. Role of folic acid depletion on homocysteine serum level in children and adolescents with epilepsy and different MTHFR C677T genotypes. Seizure. 2012 Jun;21(5):340-3. doi: 10.1016/j.seizure.2012.02.011. Epub 2012 Mar 16. PMID 22425007
- [Background] Linnebank M, Moskau S, Semmler A, Widman G, Stoffel-Wagner B, Weller M, Elger CE. Antiepileptic drugs interact with folate and vitamin B12 serum levels. Ann Neurol. 2011 Feb;69(2):352-9. doi: 10.1002/ana.22229. Epub 2011 Jan 19. PMID 21246600
- [Background] De Lourdes Levy M, Larcher V, Kurz R; Ethics Working Group of the Confederation of European Specialists in Paediatrics (CESP). Informed consent/assent in children. Statement of the Ethics Working Group of the Confederation of European Specialists in Paediatrics (CESP). Eur J Pediatr. 2003 Sep;162(9):629-33. doi: 10.1007/s00431-003-1193-z. Epub 2003 Jul 19. PMID 12884032
- [Background] Age limits and adolescents. Paediatr Child Health. 2003 Nov;8(9):577-8. doi: 10.1093/pch/8.9.577. No abstract available. PMID 20019831
- See also: World Health Organization. [Accessed May 15, 2014]; Health topics. Adolescent health. 2011 — http://www.who.int/topics/adolescent_health/en/